CLINICAL TRIAL: NCT06177093
Title: A Pilot Study of Dose dE-eScalaTion IN prostATe radIOtherapy usiNg the MRL
Brief Title: De-escalated Dose SBRT in Localized Prostate Cancer (DESTINATION-MRL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DESTINATION-MRL
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Newly diagnosed intermediate risk localized prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single centre phase II non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): All radiotherapy will be delivered on the MR-linac
  Interventions: Radiation: MR Linac delivered Radiotherapy

INTERVENTIONS:
Radiation: MR Linac delivered Radiotherapy — All radiotherapy will be delivered on the MR-linac. The whole prostate will receive 30 Gy in 5 fractions and the dominant lesion plus intra-prostatic margin will receive an isotoxic 45 Gy prescription.

SUMMARY:
This study is a single centre feasibility trial. The trial will recruit men with intermediate risk localised prostate cancer who will all receive targeted dose (escalated/de-escalated dose directed by MRI) 5 fraction SBRT to the prostate.

Trial Objectives are:

1. Primary To develop a 5 fraction de-escalated dose SBRT protocol capable of reducing side effects
2. Secondary

   * To assess levels of acute GU and GI toxicity (CTCAE)
   * To assess levels of late GU and GI toxicity (CTCAE)
   * To assess late sexual quality of life (expanded EPIC, IIEF-5)
   * To assess biochemical relapse-free survival at 2

DETAILED DESCRIPTION:
TRIAL POPULATION: Men with intermediate risk localized prostate cancer TRIAL TREATMENT: All radiotherapy will be delivered on the MR-linac. Intraprostatic dose will be varied according to risk of local recurrence, based on mpMRI, PSA and histology. The whole prostate will receive 30 Gy in 5 fractions and the dominant lesion plus intra-prostatic margin will receive an isotoxic 45 Gy prescription.

Study rationale: The DESTINATION project aims to establish whether focusing radiation dose on the area most at risk of recurrence, and reducing the dose elsewhere, can produce a low level of side effects and maximize quality of life. This trial will assess technical feasibility of this approach.

TRIAL DESIGN: DESTINATION is run as a single centre trial embedded within the Sunnybrook REB approved MOMENTUM collaboration. The MOMENTUM trial facilitates data sharing across participating institutes.

Patients will be reviewed and complete toxicity assessments (CTCAE version 5) at the end of their radiation and then at 4 and 12 weeks after completion of treatment. They will thereafter be assessed at 6, 12 and 24 months with CTCAE version 5 and the patient reported IPSS assessment completed at each time point. Thereafter follow up will be as per standard care. Patient reported EPIC-26 will be measured at; baseline, 4 and 12 weeks, and 6, 12 and 24 months from the end of radiotherapy. IIEF-5 will be completed at months 6, 12 and 24. Scans will be taken before and during radiotherapy on the MR-linac. Patients will be followed up for recurrence/biochemical failure on protocol for 24 months and thereafter as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥18 years
* Histological confirmation of prostate adenocarcinoma requiring radical radiotherapy
* Gleason score 3+3, 3+4 or 4+3 (Grade groups 1, 2 or 3)
* MRI stage T2 or less (as staged by AJCC TNM 2018)
* MRI-visible tumour(s) of PIRADS v2 grade 3 or higher on T2 and diffusion-weighted imaging and/or dynamic contrast-enhanced imaging (multiparametric MRI or mpMRI) with concordant pathology
* Tumour nodule visible on MRI occupying <50% of prostate on any axial slice and <50% prostate volume
* PSA <20 ng/ml prior to starting ADT (if applicable)
* Short course (< 6 months) concurrent androgen deprivation therapy (antiandrogens or LHRH analogues) allowed though not mandated as per the discretion of the treating physician.
* WHO Performance status 0-2
* Ability of the participant understand and the willingness to sign a written informed consent form.
* Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

* Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
* IPSS 19 or higher
* High grade disease (GG3) occult to MRI-defined lesion
* Post-void residual >100 mls, where known
* Prostate volume >90cc
* Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
* Unilateral or bilateral total hip replacement, or other pelvic metalwork which causes artefact on diffusion-weighted imaging
* Previous pelvic radiotherapy
* Patients needing >6 months of ADT due to disease parameters as per the discretion of the treating physician
* Previous invasive malignancy within the last 2 years excluding basal or squamous cell carcinomas of the skin, low risk non-muscle invasive bladder cancer (assuming cystoscopic follow up now negative) or small renal masses on surveillance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with prostate cancer
Enrollment: 20 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical Feasibility | 4 years
  To establish the technical feasibility of treating prostate cancer with toxicity-minimising. radiotherapy on an MR-linac. Patients will be followed up for recurrence/biochemical failure as per standard care.

SECONDARY OUTCOMES:
Acute and Late Toxicities | Upto 2 years post treatment
  CTCAE Version 5

CONTACTS AND LOCATIONS:
Overall Officials: Danny Vesprini, M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338